CLINICAL TRIAL: NCT01205750
Title: Basal and Insulin Mediated VLDL-triglyceride Kinetics in Obesity; Relationship With Hepatic Insulin Sensitivity
Brief Title: Hepatic Insulin Sensitivity and Very Low Density Lipoprotein Triglyceride (VLDL-TG) Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Søren Nielsen, DMSc, Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Denmark
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-0132
Record Dates: First submitted 2010-08-24; First posted 2010-09-20 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Obesity; Dyslipidemia
MeSH Terms: conditions — Obesity; Dyslipidemias | interventions — Glucose Clamp Technique; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucose clamp (Experimental)
  Interventions: Other: Glucose clamp

INTERVENTIONS:
Other: Glucose clamp — 450 min hyperinsulinemic euglycemic glucose clamp, 0,5 mU / kg lean body mass / min
  Other Names: Human insulin

SUMMARY:
Obesity is associated with dyslipidemia, which is a major risk factor for coronary heart disease. Triglycerides (TG) and cholesterol are transported in the system of lipoproteins, and the metabolism of these lipids in plasma is closely interrelated. Evidence suggests that increased concentration of very low-density lipoprotein triglyceride (VLDL-TG) is a central pathophysiological feature of the lipid and lipoprotein abnormalities in dyslipidemia.

The primary objective of this study is to investigate VLDL-TG kinetics and hepatic insulin sensitivity in age-matched obese and lean, healthy men in the postabsorptive state and during acute hyperinsulinemia using VLDL-TG and glucose tracers.

DETAILED DESCRIPTION:
Extensive description not included.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI < 25 kg/m2 or > 30 kg/m2
* Informed consent

Exclusion Criteria:

* Alcohol misuse
* Smoking
* Use of prescription drugs

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
VLDL-TG kinetics | VLDL-TG kinetics are determined postabsorptively (250 minues) and during acute hyperinsulinemia (450 minutes)
  VLDL-TG secretion rates(umol/min) and clearance rates (ml/min)are determined during 30 min steady state periods postabsorptively and using acute hyperinsulinemia using primed-constant infusion of ex vivo-labelled 14C-VLDL-TG tracer and traditional tracer dilution technique.

SECONDARY OUTCOMES:
Hepatic insulin sensitivity | Glucose kinetics are determined postabsorptively (250 minues) and during acute hyperinsulinemia (450 minutes)
  Hepatic glucose production (mg/min) is determined during 30 min steady state periods postabsorptively and during acute hyperinsulinemia using primed constant infusion og 3H-glucose tracer and traditional tracer dilution technique.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Nielsen, DMSc, Principal Investigator — Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Denmark
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark